CLINICAL TRIAL: NCT06996509
Title: Prospective, Randomized, Controlled, Open-Label Single-Center Trial Comparing High-Velocity Nasal Insufflation (HVNI) Versus Non-Invasive Ventilation (NIV) for Acute Respiratory Failure in Guillain-Barré Syndrome
Brief Title: Noninvasive Support for Acute Respiratory Failure in Guillain-Barré Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Shaddad, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 237890-5-2025
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Guillain-Barre Syndrome
Keywords: GBS
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The study employs a parallel assignment model with randomized allocation in an open-label design. In this framework, participants are prospectively assigned by chance to one of two concurrent intervention arms and remain in that arm throughout the trial. At the same time, both investigators and patients are aware of the assigned treatment. This arrangement improves the trustworthiness of the results by avoiding any leftover effects from earlier treatments, ensures that the groups are similar for comparison by randomly choosing participants, and makes it easier to provide quick respiratory support for Guillain-Barré syndrome.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blinding involves masking only those individuals who measure or adjudicate study endpoints, while participants and treating clinicians remain aware of treatment allocation. This approach reduces detection bias in outcome measurement without the logistical challenges of fully double-blinded designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Invasive Ventilation (NIV) (Experimental): Device & Settings
  Bi-level positive airway pressure (BiPAP) is set with an inspiratory positive airway pressure (IPAP) of 10-16 cmH₂O and an expiratory positive airway pressure (EPAP) of 5-8 cmH₂O.
  Adjust the fraction of inspired oxygen (FiO₂) to achieve an oxygen saturation (SpO₂) of ≥ 92%.
  Interventions: Device: Non-Invasive Ventilation (NIV)
- High velocity nasal insufflation (HVNI) (Experimental): Device & Settings
  The high-velocity nasal cannula system delivers heated, humidified gas at flow rates of 35-60 L/min.
  FiO₂ titrated to maintain SpO₂ ≥ 92 %.
  Interventions: Device: High Velocity Nasal Insufflation

INTERVENTIONS:
Device: Non-Invasive Ventilation (NIV) — Bi-Level NIV delivers two preset pressure levels-Inspiratory Positive Airway Pressure (IPAP) and Expiratory Positive Airway Pressure (EPAP)-via a tightly fitting mask interface
  Other Names: Bi-level Positive airway pressure ventilation (BIPAP)
  Arms: Non-Invasive Ventilation (NIV)
Device: High Velocity Nasal Insufflation — High-Velocity Nasal Cannula therapy delivers heated, humidified gas at flow rates exceeding patients' peak inspiratory demands (35-60 L/min), with precise FiO₂ control up to 100 %
  Other Names: High velocity nasal cannula; Vapotherm Delivery system
  Arms: High velocity nasal insufflation (HVNI)

SUMMARY:
This study will involve 70 adult patients with Guillain-Barré syndrome who have severe breathing problems. It will compare two types of breathing support: high-velocity nasal cannula (HVNC) (which delivers heated and humidified air at 35-60 L/min) and bi-level noninvasive ventilation (NIV) (which uses two pressure levels: inspiratory positive airway pressure (IPAP) 10-16 cmH₂O and expiratory positive airway pressure (EPAP) 5-8O). The main goal is to see how many patients can stop using non-invasive support without needing a breathing machine by Day 30. Other goals include how long it takes to stop using support, how comfortable patients feel, how long they stay in the ICU or hospital, how many days they can breathe on their own, and the number of deaths in 30 days. The main goal is to see how many patients can stop using non-invasive support without needing invasive ventilation by Day 30, while also looking at other factors like how long it takes to stop assistance, how comfortable patients are, how long they stay in the hospital, how many days they can breathe on their own, the number of deaths within 30 days, and their overall health.

DETAILED DESCRIPTION:
Guillain-Barré Syndrome (GBS) is an acute autoimmune disorder characterized by rapid-onset muscle weakness due to peripheral nerve damage. A significant complication in GBS is respiratory failure, occurring in approximately 25% of cases, necessitating timely and effective respiratory support to prevent morbidity and mortality.

Non-invasive ventilation (NIV) is a standard intervention for managing acute respiratory failure, particularly in conditions such as chronic obstructive pulmonary disease (COPD). NIV delivers positive pressure ventilation through interfaces such as oronasal masks, providing support without the need for endotracheal intubation. While effective, NIV can be associated with patient discomfort, skin breakdown, and challenges in secretion management, potentially leading to intolerance or failure of the therapy.

High-flow nasal cannula (HFNC) therapy has emerged as an alternative respiratory support modality. HFNC delivers heated and humidified oxygen at high flow rates through nasal prongs, offering several physiological benefits:

Enhanced Oxygenation: By delivering high flow rates, HFNC can meet or exceed the patient's inspiratory demand, ensuring consistent oxygen delivery.

Reduction in Work of Breathing: The continuous flow can generate a low level of positive airway pressure, decreasing the effort required for breathing.

Enhanced Secretion Clearance: Humidified gas supports mucociliary function, facilitating the clearance of secretions.

Patient Comfort: The nasal interface is generally better tolerated than masks used in non-invasive ventilation (NIV), potentially improving adherence to therapy.

Recent studies have explored the efficacy of HFNC compared to NIV in various forms of respiratory failure. While NIV remains the first-line treatment in many scenarios, HFNC has shown promise in improving patient comfort and reducing the need for escalation to invasive mechanical ventilation in specific patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* GBS per Brighton criteria (clinical ± cerebrospinal fluid (CSF)/electrodiagnostics)
* Moderate acute respiratory failure (vital capacity (VC) 15-20 mL/kg and/or arterial partial pressure of carbon dioxide (PaCO₂) > 45 mmHg or arterial partial pressure of oxygen (PaO₂) < 70 mmHg on room air (RA) and/or respiratory rate (RR) > 24 /min)
* Hughes Grade 3-4, The Erasmus Guillain-Barré Syndrome Respiratory Insufficiency Score (EGRIS) 1-3, Medical Research Council (MRC) sum score 20-40
* Glasgow Coma Scale (GCS) ≥ 13, intact cough/gag, stable hemodynamics
* Onset of respiratory symptoms ≤ 7 days

Exclusion Criteria:

* Chronic respiratory disease (COPD, interstitial lung diseases (ILD), persistent asthma)
* Immediate need for invasive ventilation (VC < 10 mL/kg, unresponsive severe gas-exchange derangement)
* Severe bulbar dysfunction or prior intubation for the current illness
* Contraindications to HVNC/NIV (facial trauma, untreated pneumothorax, agitation, vomiting)
* Pregnancy
* Severe comorbidity limiting prognosis.
* Declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximize the successful weaning duration in days. | 48 hours after randomization and daily for 28 days.
  Examine and compare the percentage of Guillain-Barré syndrome patients who can discontinue using their assigned non-invasive support (HVNC or NIV) without requiring a switch to invasive mechanical ventilation during their initial stay in the intensive care unit (ICU), which will be from 48 hours of randomization and daily for 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Shaddad, MD, Principal Investigator — Assiut University; Aliae A. Hussien, MD, Principal Investigator — Assiut University
Locations (1):
- Assuit Univeristy, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data supporting the primary and secondary outcomes, along with accompanying data dictionaries and the statistical analysis plan, will be made available by Assiut University's institutional data-sharing policies. Data will be accessible 6-36 months after publication to qualified researchers upon submission of a study proposal, approval by the University Research Ethics Committee, and execution of a data-use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: 6-36 months after publication
Access Criteria: Qualified researchers must submit a study proposal, obtain approval from the University Research Ethics Committee, and execute a data-use agreement.